CLINICAL TRIAL: NCT06174753
Title: The University of Ottawa Dapagliflozin in STEMI Randomized Clinical Trial
Brief Title: Dapagliflozin in STEMI
Acronym: DAPA STEMI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230332-01H
Record Dates: First submitted 2023-12-07; First posted 2023-12-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: ST Elevation Myocardial Infarction; Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: a single center, randomized, double-blind, parallel group study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Dapagliflozin 10mg daily X 7 days
  Interventions: Drug: Dapagliflozin 10mg Tab; Diagnostic Test: CMR
- Placebo (Placebo Comparator): Placebo daily X 7 days
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg daily X 7 days
  Arms: Treatment
Diagnostic Test: CMR — CMR 3-5 days post randomization

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of SGLT2i in limiting infarct size in patients with STEMI referred for PPCI.

Eligible STEMI patients enrolled into the trial will be randomized to a SGLT2i or placebo.

Cardiovascular Magnetic Resonance (CMR) imaging will be used to determine the infarct size.

DETAILED DESCRIPTION:
DAPA STEMI is a single center, randomized, double-blind, parallel group study in which eligible participants with a STEMI and undergoing PPCI will be recruited and randomly assigned to dapagliflozin or placebo to take for 7 days. Participants will be prescribed study treatment i.e. dapagliflozin (10 mg) or placebo daily for 7 days.

A CMR will be obtained at day 3-5 to assess for infarct size. Participants will have follow-up visits at 30, 90, and 180 days to assess for cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

Patients referred for PPCI meeting the following criteria are eligible for the study:

* Ischemic chest discomfort of ≥30 minutes duration, and
* Onset of chest pain ≤12 hours prior to entry into the study, and
* One of the following High-Risk criteria on a standard 12 lead ECG:

  a. Anterior STEMI with ST-segment elevation ≥2mm (0.2 mV) in each of at least 2 contiguous precordial leads (V1-V6) b. Extensive non-anterior STEMI defined as ST-segment elevation of >1mm in two or more contiguous non-anterior leads accompanied by i. 8 or more leads with > 1 mm ST elevation or depression, or both; OR ii. Sum of ST- segment elevation >20mm

Exclusion Criteria:

* Age < 18 years
* Any contraindication to undergo CMR imaging
* Killip 4 (Cardiogenic shock on presentation)
* Therapy with SGLT2i within last 8 weeks
* Type 1 diabetes mellitus
* Pregnancy
* Nursing mother
* Unwilling to use appropriate forms of contraception, as applicable
* Chronic symptomatic HF with prior hospitalization for HF within the last year
* hospitalization
* Known history of prior MI
* Any non-CV condition with a life expectancy of less than one year
* Previous randomization in the present study
* Participation in a study with another investigational device or drug < four weeks
* Inability to provide informed consent
* Confirmed ketoacidosis at time of admission
* Known severe hepatic impairment (Cirrhosis)
* Severe renal impairment (eGFR < 30 mL/min1.73m2 (based on prior or baseline blood work)
* Known severe valvular heart disease
* Need for CABG within 90 days based on the results of the initial coronary angiogram
* False positive STEMI (based on the results of the coronary angiogram)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Infarct Size | 3-5 days
  Infarct size (% of total LV mass) measured by CMR

SECONDARY OUTCOMES:
Incidence of Multiple Cardiac Adverse Events (MACE) | 3 months, and 6 months
  A composite of death, reinfarction, stroke, or rehospitalization for HF
Number of participants with Cardiogenic Shock | during initial hospitalization (*up to 30 days)
  Evaluated using the SCAI classification; only class C, D, or E will be adjudicated as a secondary outcome
Number of Participants with Acute Kidney Injury | 3 months, and 6 months
  As defined according to the KDIGO definition

CONTACTS AND LOCATIONS:
Overall Officials: Michel LeMay, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No